CLINICAL TRIAL: NCT05927857
Title: A Phase Ib/II Study of Ramucirumab (Cyramza®), Nal-IRI (ONIVYDE®) and Trifluridine/Tipiracil (Lonsurf®) in Second Line Metastatic Gastric Cancer (COOL Study).
Brief Title: Ramucirumab (Cyramza), Nal-IRI (ONIVYDE) and Trifluridine/Tipiracil (Lonsurf) in Second Line Metastatic Gastric Cancer .
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1223
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Gastric Adenocarcinoma; Second Line; Chemotherapy
Keywords: nal-IRI (ONIVYDE); TAS-102 (LONSURF); Ramucirumab (Cyramza)
MeSH Terms: interventions — irinotecan sucrosofate; Ramucirumab; Trifluridine; tipiracil; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 1b/II (Experimental): * Infusional nal-IRI (ONIVYDE, free form) 50/60/70 mg/m2 over 90 minutes day 1.
  * Infusional Ramucirumab(Cyramza)8 mg/kg over 60 minutes day 1.
  * oral Trifluridine/Tipiracil TAS-102 (LONSURF) 30 mg/m2/b.i.d. day 1-5.
  * Every 14 days count as one cycle.
  Interventions: Drug: nal-IRI /Experimental; Drug: Ramucirumab /Experimental; Drug: Trifluridine/Tipiracil /Experimental

INTERVENTIONS:
Drug: nal-IRI /Experimental — infusional 50/60/70 mg/m2 over 90 minutes day 1, every 14 days.
  Other Names: ONIVYDE
Drug: Ramucirumab /Experimental — infusional 8mg/kg over 60 minutes day 1, every 14 days.
  Other Names: Cyramza
Drug: Trifluridine/Tipiracil /Experimental — oral 30 mg/m2/b.i.d. day 1-5, every 14 days.
  Other Names: LONSURF

SUMMARY:
Primary Objectives

* In phase 1b cohort, to determine MTD (maximum tolerated dose) of nal-IRI (ONIVYDE®) in combination with Ramucirumab (Cyramza®) and TAS-102 (LONSURF®)
* In phase II cohort, to evaluate disease objective response rate (ORR) of Ramucirumab (Cyramza®), nal-IRI (ONIVYDE®) in combination with TAS-102 (LONSURF®) Secondary Objectives
* To evaluate disease control rate (DCR)
* To evaluate progression-free survival (PFS)
* To evaluate overall survival (OS)
* To assess the safety profile
* To study the blood biomarkers

DETAILED DESCRIPTION:
* Eligible patients will be treated with infusional nal-IRI (ONIVYDE®, free form) 50/60/70 mg/m2 over 90 minutes day 1, Ramucirumab 8 mg/kg over 60 minutes day 1, in combination with oral TAS-102 (LONSURF®) 30 mg/m2/b.i.d. day 1-5, every 14 days.
* Every 14 days count as one cycle.
* Patients will be treated until disease progression, unacceptable toxicity or other condition meeting the off-study criteria.
* Scheme of phase 1b: dose Level 0 to 2 will be tested with the following dose levels:
* Dose level 0= Ramucirumab(Cyramza®) 8mg/kg on day 1, nal-IRI (ONIVYDE®, free form) 50 mg/m2 on day 1 plus Trifluridine/Tipiracil (Lonsurf®) 30mg/m2 on day 1-5, q2wk
* Dose level 1= Ramucirumab(Cyramza®) 8mg/kg on day 1, nal-IRI (ONIVYDE®, free form) 60 mg/m2 on day 1 plus Trifluridine/Tipiracil (Lonsurf®) 30mg/m2 on day 1-5, q2wk
* Dose level 2= Ramucirumab(Cyramza®) 8mg/kg on day 1, nal-IRI (ONIVYDE®, free form) 70 mg/m2 on day 1 plus Trifluridine/Tipiracil (Lonsurf®) 30mg/m2 on day 1-5, q2wk
* Adaptive phase IB cohort:
* 3+3 dose escalation will be applied for phase Ib cohort. All treated patients of MTD dose level in phase 1b cohort will be incorporated into phase II cohort for final analysis. No intra-patient dose escalation is allowed during DLT period. Patients could only have dose modification after the DLT period. G-CSF prophylaxis is not allowed in DLT period.
* Dose escalation rule: Two to six patients will be enrolled in each cohort depending on cases with DLTs. The starting dose is dose level 0. If none of the first 3 patients experiences DLT, then dose escalation will proceed to the next cohort of patients. If only 1 of 3 patients developed DLT, the cohort will be expanded to 6 patients. If more than 1 patient developed DLT at a certain dose level/group, the dose level/group is considered intolerable to the patients. If no more than 1 out of 6 patients experience DLT, the dose level/group is considered tolerable. A minimum of 6 evaluable patients will be treated at the MTD. The MTD at which no more than 1 of the 6 patients experience DLT will be determined for the phase II cohort. Based on results from phase IB cohort, MTD will be determined. All treated population in MTD cohort will be incorporated into phase II cohort for final analysis.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically confirmed metastatic gastric adenocarcinoma
2. patients have received only first line of systemic therapy, including recurrence during adjuvant therapy or within 6 months after the completion of adjuvant treatment.
3. ECOG(Eastern Cooperative Oncology Group) performance status 0 or 1
4. patients with HER2/neu-positive tumor must be exposure to Herceptin treatment
5. at least one measurable disease according to the RECIST version 1.1;
6. patients are aged 20 to 80 years;
7. patients have a life expectancy ≥ 3 months;
8. patients have adequate renal function with defined as serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or Ccr ≥ 40 mL/min;
9. patients with adequate hepatic function as defined by a total bilirubin ≤1.5 times the ULN, and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times the ULN or 5 times the ULN in the setting of liver metastases.
10. patients have adequate bone marrow function, defined as an absolute neutrophil count ≥ 1500/mm3, hemoglobin ≥9 g/dL, and platelet count ≥ 100,000/mm3 (transfusion or G-CSF support before enrollment is allowed)
11. patients have International Normalized Ratio (INR) ≤1.5 and a partial thromboplastin time (PTT) (PTT/aPTT) < 1.5 x ULN;
12. patients' urinary protein is ≤1+ on dipstick or routine urinalysis or a 24-hour urine collection for protein must demonstrate <1000 mg of protein if urine dipstick or routine analysis is ≥ 2+;
13. patients with childbearing potential shall have effective contraception for both the patient and his or her partner during the study;
14. female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to first dose of protocol therapy;
15. the ability to understand and willingness and to sign a written informed consent document.

Exclusion Criteria:

1. patient can't take oral drugs;
2. known hypersensitivity to irinotecan, fluoropyrimidine, or ramucirumab;
3. receipt of surgery within the past 4 weeks before study enrollment;
4. ≥ grade 2 diarrhea and ascites
5. concurrent severe infection with intravenous systemic antibiotics treatment;
6. patients have experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy;
7. patients have a prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation;
8. patients have:

   * cirrhosis at a level of Child-Pugh B (or worse) or
   * cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis;
9. patients have a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy;
10. patients have undergone major surgery within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to the first dose of protocol therapy. Patients have elective or planned major surgery to be performed during the course of the clinical trial;
11. patients have uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management;
12. patients have experienced any grade 3-4 GI bleeding within 3 months prior to first dose of protocol therapy;
13. patients have a history of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy;
14. patients are receiving chronic antiplatelet therapy, including dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted;
15. previously received prior nal-IRI (ONIVYDE®) or TAS-102 (LONSURF®) or ramucirumab therapy
16. another previous malignancy diagnosed within the past 5 years except for non melanoma skin cancer or stage I cervical cancer;
17. pregnant or breast feeding women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine MTD (maximum tolerated dose) of nal-IRI (ONIVYDE) | Phase I last patient in has been treated for 28 days.
  All treated patients of MTD dose level in phase 1b cohort will be incorporated into phase II cohort for final analysis.
To evaluate disease objective response rate (ORR) | Whichever occurs first assessed up to 24 months.
  Based on results from phase Ib cohort, MTD will be determined. All treated population in MTD cohort will be incorporated into phase II cohort for final analysis.

SECONDARY OUTCOMES:
•To evaluate disease control rate (DCR) | The time from registration to death from any cause assessed up to 24 months.
  •Patients will be treated until disease progression, unacceptable toxicity or other condition meeting the off-study criteria.
•To evaluate progression-free survival (PFS) | The time from registration to occurrence of progression based on the tumor response assessment by scheduled or un- scheduled CT scan or MRI. (whichever occurs first assessed up to 24 months)
  • objective tumor response according to RECIST v1.1 guidelines.
•To evaluate overall survival (OS) | The time from registration to death from any cause assessed up to 24 months.
  the time from the date of first study treatment to the date of patient death, due to any cause, or to the last date the patient was known to be alive.
•To assess the safety profile | The time from registration to death from every 14 days assessed up to 24 months.
  •Safety evaluations: physical examination, vital signs, body weight, ECOG performance status, clinical laboratory values (biochemistry, hematology, and urinalysis), and any adverse event (AE) graded by using CTCAE v5.0 if applicable.
•To study the blood biomarkers | The time from baseline on day 1.
  * To evaluate the drug sensitivity of circulating tumor cells to, including but not limited to irinotecan, fluorouracil and ramucirumab.
  * Patients enrolled in both phase Ib and phase II parts will participate in biomarker study

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Jung Chiang, MD-PhD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan/Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Innocenti F, Kroetz DL, Schuetz E, Dolan ME, Ramirez J, Relling M, Chen P, Das S, Rosner GL, Ratain MJ. Comprehensive pharmacogenetic analysis of irinotecan neutropenia and pharmacokinetics. J Clin Oncol. 2009 Jun 1;27(16):2604-14. doi: 10.1200/JCO.2008.20.6300. Epub 2009 Apr 6. PMID 19349540
- [Result] Mathijssen RH, van Alphen RJ, Verweij J, Loos WJ, Nooter K, Stoter G, Sparreboom A. Clinical pharmacokinetics and metabolism of irinotecan (CPT-11). Clin Cancer Res. 2001 Aug;7(8):2182-94. PMID 11489791
- [Result] Smith NF, Figg WD, Sparreboom A. Pharmacogenetics of irinotecan metabolism and transport: an update. Toxicol In Vitro. 2006 Mar;20(2):163-75. doi: 10.1016/j.tiv.2005.06.045. Epub 2005 Nov 3. PMID 16271446
- [Result] Kawato Y, Aonuma M, Hirota Y, Kuga H, Sato K. Intracellular roles of SN-38, a metabolite of the camptothecin derivative CPT-11, in the antitumor effect of CPT-11. Cancer Res. 1991 Aug 15;51(16):4187-91. PMID 1651156
- [Result] Garcia-Carbonero R, Supko JG. Current perspectives on the clinical experience, pharmacology, and continued development of the camptothecins. Clin Cancer Res. 2002 Mar;8(3):641-61. PMID 11895891
- [Result] Vanhoefer U, Harstrick A, Achterrath W, Cao S, Seeber S, Rustum YM. Irinotecan in the treatment of colorectal cancer: clinical overview. J Clin Oncol. 2001 Mar 1;19(5):1501-18. doi: 10.1200/JCO.2001.19.5.1501. PMID 11230497
- [Result] Lee DH, Kim HT, Han JY, Lee SY, Yoon SJ, Kim HY, Lee JS. A phase II trial of modified weekly irinotecan and cisplatin for chemotherapy-naive patients with metastatic or recurrent squamous cell carcinoma of the esophagus. Cancer Chemother Pharmacol. 2008 Jan;61(1):83-8. doi: 10.1007/s00280-007-0450-7. Epub 2007 Apr 28. PMID 17468871
- [Result] Chen SC, Chang PM, Yang MH. Cisplatin/Tegafur/Uracil/Irinotecan Triple Combination Therapy for Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma: A Phase I/II Clinical Study. Oncologist. 2016 May;21(5):537-8. doi: 10.1634/theoncologist.2015-0515. Epub 2016 Apr 18. PMID 27091418
- [Result] Tsai CS, Park JW, Chen LT. Nanovector-based therapies in advanced pancreatic cancer. J Gastrointest Oncol. 2011 Sep;2(3):185-94. doi: 10.3978/j.issn.2078-6891.2011.034. PMID 22811849
- [Result] Chang TC, Shiah HS, Yang CH, Yeh KH, Cheng AL, Shen BN, Wang YW, Yeh CG, Chiang NJ, Chang JY, Chen LT. Phase I study of nanoliposomal irinotecan (PEP02) in advanced solid tumor patients. Cancer Chemother Pharmacol. 2015 Mar;75(3):579-86. doi: 10.1007/s00280-014-2671-x. Epub 2015 Jan 11. PMID 25577133
- [Result] Chiang NJ, Chao TY, Hsieh RK, Wang CH, Wang YW, Yeh CG, Chen LT. A phase I dose-escalation study of PEP02 (irinotecan liposome injection) in combination with 5-fluorouracil and leucovorin in advanced solid tumors. BMC Cancer. 2016 Nov 21;16(1):907. doi: 10.1186/s12885-016-2933-6. PMID 27871319
- [Result] Roy AC, Park SR, Cunningham D, Kang YK, Chao Y, Chen LT, Rees C, Lim HY, Tabernero J, Ramos FJ, Kujundzic M, Cardic MB, Yeh CG, de Gramont A. A randomized phase II study of PEP02 (MM-398), irinotecan or docetaxel as a second-line therapy in patients with locally advanced or metastatic gastric or gastro-oesophageal junction adenocarcinoma. Ann Oncol. 2013 Jun;24(6):1567-73. doi: 10.1093/annonc/mdt002. Epub 2013 Feb 13. PMID 23406728
- [Result] Ko AH, Tempero MA, Shan YS, Su WC, Lin YL, Dito E, Ong A, Wang YW, Yeh CG, Chen LT. A multinational phase 2 study of nanoliposomal irinotecan sucrosofate (PEP02, MM-398) for patients with gemcitabine-refractory metastatic pancreatic cancer. Br J Cancer. 2013 Aug 20;109(4):920-5. doi: 10.1038/bjc.2013.408. Epub 2013 Jul 23. PMID 23880820
- [Result] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328